CLINICAL TRIAL: NCT01059123
Title: Randomized Non Inferiority Study Comparing Short Course of Oral Amoxicillin to One of the Usual Treatments of Lower Leg Erysipelas
Brief Title: Short Course of Amoxicillin for Erysipelas
Acronym: SHARE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient number of inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government); Société de Dermatologie Française (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P071207; 2008-006794-32 (EudraCT Number)
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Erysipelas
Keywords: Amoxicillin; Erysipelas; Short course
MeSH Terms: conditions — Erysipelas | interventions — Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1:Short treatment (Experimental): amoxicillin ; 50 mg/kg/24H ; P.O. ; 3 times/day 6 days.
  Interventions: Drug: Amoxicillin
- 2:Usual treatment (Active Comparator): amoxicillin 50 mg/kg/24H ; I.V. ; 3 times/day ; up to apyrexia then amoxicillin ; 50 mg/kg/24H ; P.O. ; 3 times/day up to day 14.
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — 50 mg/kg/24H ; Per Os ; 3 times/day 6 days
  Arms: 1:Short treatment
Drug: Amoxicillin — 50 mg/kg/24H in I.V. ; 3 times/day ; up to apyrexia then amoxicillin ; 50 mg/kg/24H ; Per Os ; 3 times/day up to day 14.
  Arms: 2:Usual treatment

SUMMARY:
The propose of this study is to determine whether a 6-day duration of oral amoxicillin treatment of erysipelas is non-inferior to a 14-day standard duration intravenous then oral amoxicillin regimen. This trial will be open but evaluation will be perform by a blind evaluator.

DETAILED DESCRIPTION:
To fight against increasing rate of bacterial resistance to antibiotics, several studies have demonstrated efficacy of short antibiotic course in e.g. acute streptococcal tonsillitis, community acquired pneumonia, and urinary tract infection. Erysipelas is an acute dermo-hypodermal infection due to streptococcus. To date no resistance of theses bacteria to amoxicillin was described. The diagnosis of erysipelas is clinical. Thus, short course of antibiotic is a good regimen to test in erysipelas treatment. To date there is no controlled trial concerning efficacy of oral amoxicillin in erysipelas treatment. Expected advantages of the demonstration of the non inferiority of a short and oral amoxicillin treatment in erysipelas are: reduction of antibiotic selective pressure, cost, adverse events caused by infusion and hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* First episode of erysipelas of a lower leg defined as

  * acute well delineate inflammation than had lasted less than 5 days
  * T°≥ 38°5 at least once during the past 5 days or chills.
  * Score ≥3 : oedema, erythema, pain each scored from 0 to 3 : 0= none, 1= moderate, 3= severe
* Written informed consent provided by the patient
* available health insurance
* accept conditions of the trial

Exclusion Criteria:

* Erysipelas for more than 5 days
* Score < 3
* Septic shock
* Clinical signs of necrotizing cellulitis or fasciitis, bullous lesions related to necrosis, purpuric lesions or superficial cutaneous necrosis.
* Past history of erysipelas of the same lower leg
* Erysipelas not on the lower leg
* Bilateral erysipelas
* Bite occuring during the preceding 7 days.
* Diabetic foot
* patients who have previously received systemic antibiotherapy within the last 5 days (except one or two doses within last 24 hours)
* History of any hypersensitivity or allergic reaction to beta-lactam drugs
* Known renal or Hepatic failure
* Known HIV infection
* Female patients who are pregnant, lactating (breast milk feeding), or who are of child bearing potential and not using an acceptable method of birth control
* Impossibility to stop immunosuppressive treatment, systemic corticosteroids or nonsteroidal anti-inflammatory drugs.
* Severe gastrointestinal disease, dysphagia or any pathology preventing oral administration of treatment.
* Denied to sign written informed consent
* Unable or unwilling to adhere to the study-specified procedures and restrictions
* Evolutive cancer under treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Clinical cure rate defined as body temperature ≤ 37,5°and disappearance of the cutaneous plaque (score=o) | Day 30 ± 5

SECONDARY OUTCOMES:
Time to obtain disappearance of fever and local signs | up to day 30 ± 5
Relapse rate | end of treatment to day 30± 5
Recurrence rate | day 30± 5 to day 95± 5
Frequency of adverse events | 30 days ± 5

CONTACTS AND LOCATIONS:
Overall Officials: Olivier CHOSIDOW, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Henri Mondor - Service de dermatologie, Créteil, Île-de-France Region, France